CLINICAL TRIAL: NCT03535298
Title: Determining the Effectiveness of earLy Intensive Versus Escalation Approaches for the Treatment of Relapsing-Remitting Multiple Sclerosis
Brief Title: Determining the Effectiveness of earLy Intensive Versus Escalation Approaches for RRMS
Acronym: DELIVER-MS
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: University of Nottingham (Other)
Responsible Party: Principal Investigator, Daniel Ontaneda, MD, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCF 18-326/23-453
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Alemtuzumab; ocrelizumab; Natalizumab; Rituximab; ofatumumab; ublituximab; Interferon beta-1b; Interferon-beta; Glatiramer Acetate; teriflunomide; Fingolimod Hydrochloride; Coat Protein Complex I; peginterferon beta-1a; Interferon beta-1a; Dimethyl Fumarate; Cladribine; siponimod; diroximel fumarate; ozanimod; monomethyl fumarate; ponesimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- EHT: Early Highly-effective (Experimental): Participants randomized to the "EHT: Early Highly-effective" arm will receive one of the highly effective MS therapies (Ocrevus, Lemtrada, Tysabri, Rituximab, Kesimpta) as their initial disease modifying treatment.
  Interventions: one of the highly effective MS therapies
  The randomization affects only the INITIAL treatment received. Once that treatment has been initiated, any subsequent changes are made according to standard clinical practice, regardless of randomization group.
  Interventions: Drug: Early Highly Effective Therapies Group
- ESC: Escalation (Experimental): Participants randomized to the "ESC: Escalation" arm will receive any other approved MS therapy (not one of the EHT group) as their initial disease modifying treatment.
  Interventions: one of the MS therapies NOT in the highly effective group
  The randomization affects only the INITIAL treatment received. Once that treatment has been initiated, any subsequent changes are made according to standard clinical practice, regardless of randomization group.
  Interventions: Drug: Escalation Therapies Group
- OBS: Observational (No Intervention): Participants will not be restricted to a group of MS therapies.
  Participants enter this arm if they are not comfortable with randomization, are not eligible to receive any of the options in a randomized arm, or are not able to secure insurance coverage for any therapy in a randomized arm.

INTERVENTIONS:
Drug: Early Highly Effective Therapies Group — Highly Effective MS Therapy group of medications
  Other Names: Lemtrada (alemtuzumab); Ocrevus (ocrelizumab); Tysabri (natalizumab); Rituxan (rituximab); Kesimpta (ofatumumab); Briumvi (ublituximab)
  Arms: EHT: Early Highly-effective
Drug: Escalation Therapies Group — Escalation MS Therapy group of medications
  Other Names: Betaseron (beta interferon); Copaxone (glatiramer acetate); Aubagio (teriflunomide); Extavia (beta interferon); Gilenya (fingolimod); Glatopa (glatiramer acetate); Plegridy (beta interferon); Rebif (beta interferon); Tecfidera (dimethyl fumarate); Avonex (beta interferon); Mavenclad (cladribine); Mayzent (siponimod); Vumerity (diroximel fumarate); Zeposia (ozanimod); Bafiertam (monomethyl fumarate); Ponvory (ponesimod)
  Arms: ESC: Escalation

SUMMARY:
The DELIVER-MS study seeks to answer the question: Does early treatment with highly effective DMT improve the prognosis for people with MS? This is an area of significant controversy and no data currently exist to guide treatment choices for patients and clinicians. The study results will help guide overall treatment philosophy and will be applicable not only to a wide range of existing therapies but also to new therapies, meeting a significant unmet need in patient decision making and aiding the decision for medication approval by third parties.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 to 60 years.
2. Established diagnosis of MS, as defined by the 2017 revision of McDonald Diagnostic Criteria (99).
3. RRMS disease course as defined by the 2013 revisions of the MS clinical course definition (4).
4. Participants must have evidence of active disease based on: one or more MS relapses within the last 18 months prior to screening visit or radiological evidence of MS activity (≥2 new T2 lesions within the last 12 months from screening [compared to a previous recent MRI within 18 months of screening] or ≥1 GdE demonstrated on brain or spinal cord MRI performed within the last 12 months of screening).
5. Participants must be ambulatory with disease onset ≤ 5 years and treatment-naïve (i.e., no MS DMT at any time in the past).
6. Participants must be eligible to receive at least one form of DMT within each treatment arm.
7. EDSS at Baseline visit ≤ 6.5

Exclusion Criteria:

1. Participants with contraindications to all forms of DMT in either of the treatment arms.
2. Participants must never have received any of the following medications: natalizumab, alemtuzumab, ocrelizumab, rituximab, ofatumumab, cladribine, siponimod, interferon beta-1a, interferon beta-1b, pegylated interferon beta-1a, glatiramer acetate, fingolimod, teriflunomide, dimethyl fumarate, daclizumab, mitoxantrone, diroximel fumarate, ozanimod, monomethyl fumarate, ponesimod.
3. Participants must have not received any of the following medications, for reasons other than MS, in the last 12 months: cyclophosphamide, azathioprine, mycophenolate mofetil, cyclosporine, methotrexate, leflunomide, laquinimod, atacicept, other monoclonal antibodies.
4. Participants with clinically relevant medical or surgical conditions that, in the opinion of the investigator, would put the subject at risk by participating in the study
5. Participants unable to provide informed consent.
6. Contraindication or inability to undergo MRI with Gd due to metal or metal implants, allergy to Gd contrast, claustrophobia, pain, spasticity, or excessive movement related to tremor.
7. Unwillingness or inability to comply with the requirements of this protocol including the presence of any condition (physical, mental, or social) that, in the opinion of the PI, is likely to affect the participant's ability to comply with the study protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 800 (Estimated)
Dates: Start 2019-01-03 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Brain volume loss, baseline to month 36 | Baseline to 36 months
  To determine whether an EHT approach to DMT, defined as use of one of four monoclonal antibodies (alemtuzumab, natalizumab, rituximab, or ocrelizumab) as first-line therapy, is more effective than an escalation of treatment approach in reducing normalized whole brain volume loss measured using MRI in PwRRMS from Baseline to Month 36.
EDSS+, month 48 to month 108 | 48 months to 108 months
  To determine whether an EHT approach to DMT, defined as use of one of six monoclonal antibodies (alemtuzumab, natalizumab, rituximab, ocrelizumab, ofatumumab, ublituximab) as first-line therapy, is more effective than an escalation of treatment approach in reducing time to reach a multidimensional composite comprised of EDSS+ worsening. EDSS+ worsening will be defined as worsening on ⩾ 1 of the 3 components: EDSS, 9HPT, or T25FW, which is confirmed at another visit after 12 months. EDSS worsening will be defined as a ⩾1.0-point increase from a baseline score of ⩽5.5 or a ⩾0.5-point increase from a baseline score of ⩾6.0. T25FW and 9HPT worsening will be defined as ⩾20% worsening from baseline.

SECONDARY OUTCOMES:
Brain volume loss, month 6 to month 36 | Month 6 to month 36
  To determine whether an EHT approach to DMT, defined as use of one of four monoclonal antibodies (alemtuzumab, natalizumab, rituximab, or ocrelizumab) as first-line therapy, is more effective than an escalation of treatment approach in reducing normalized whole brain volume loss measured using MRI in PwRRMS from Month 6 to Month 36.
Proportion of participants with progression | Baseline to 36 months
  Proportion of participants with a multidimensional composite comprised of EDSS progression (>1.5 points for those with EDSS of 0 at Baseline, ≥1.0 for those with EDSS of 0.5-5.0 at Baseline, and >0.5 points for those with EDSS above 5.0 at Baseline), 20% change in MSFC-4 subcomponents (T25FW, 9HPT), 10% in SDMT or, 1 line change in LCLA confirmed over 12 months.
Change in MSIS-29, baseline to 36 months | Baseline to 36 months
  Change in MSIS-29 responses from participants
Change in Neuro-QOL, baseline to 36 months | Baseline to 36 months
  11 subscales, each is scored separately, there is no composite score
  Physical Domains:
  Upper Extremity Function (Fine Motor, ADL):
  Higher scores indicate: Better Functioning
  Lower Extremity Function (Mobility):
  Higher scores indicate: Better Functioning
  Fatigue:
  Higher scores indicate: Worse Functioning
  Sleep Disturbance:
  Higher scores indicate: Worse Functioning
  Mental Domains:
  Cognition Function:
  Higher scores indicate: Better Functioning
  Stigma:
  Higher scores indicate: Worse Functioning
  Anxiety:
  Higher scores indicate: Worse Functioning
  Depression:
  Higher scores indicate: Worse Functioning
  Positive Affect and Well -being:
  Higher scores indicate: Better Functioning
  Social Domains:
  Ability to Participate in Social Roles and Activities:
  Higher scores indicate: Better Functioning
  Satisfaction with Social Roles and Activities:
  Higher scores indicate: Better Functioning
Time to reach SPMS, month 48 to month 108 | 48 months to 108 months
  To determine the efficacy of an EHT approach as compared to an escalation approach as reflected by the following:
  * Time to reach secondary progressive MS (SPMS) as defined by worsening on the EDSS (3 strata definition for EDSS worsening plus EDSS score of ≥4 and pyramidal score ≥2), confirmed at 12 months, over 108 months
  * Proportion of participants with a 20% or greater change in T25FW at 108 months.
  * Proportion of participants with a 20% or greater change in 9HPT at 108 months.
  * Proportion of participants with a 20% or greater change in the SDMT at 108 months.
Efficacy difference between EHT and ESC, month 48 to month 108 | 48 months to 108 months
  To determine the efficacy of an EHT approach as compared to an escalation approach as reflected in the following patient-reported outcomes:
  * The change in participant-perceived symptoms as measured by the MSIS-29.
  * The change in participant quality of life as measured by Neuro-QOL.
Safety difference between EHT and ESC, month 48 to month 108 | 48 months to 108 months
  To determine the safety of an EHT approach as compared to an escalation approach as reflected in the following:
  * Proportion of participants with SAEs
  * Rate of SAEs
  * Proportion of participants with DMT discontinuation due to safety or tolerability concerns
  * Cumulative on-therapy TSQM Response scores

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Ontaneda, MD, MSc, Principal Investigator — The Cleveland Clinic; Nikos Evangelou, MD, DPhil, Principal Investigator — University of Nottingham
Locations (30):
- United States (15):
  - University of Colorado-Anschutz Medical Campus, Aurora, Colorado
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - University of Buffalo, Buffalo, New York
  - University Rochester Medical Center, Rochester, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio Health, Columbus, Ohio
  - UT-Austin, Austin, Texas
  - Baylor College of Medicine, Houston, Houston, Texas
  - UTHealth-Houston, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Wisconsin-Madison, Madison, Wisconsin
- United Kingdom (15):
  - University Hospitals Coventry and Warwickshire, Coventry, England
  - The Leeds Teaching Hospitals NHS Trust, Leeds General Infirmary, Leeds, England
  - University Hospitals Leicester, Leicester, England
  - Imperial College Healthcare NHS Trust, Charing Cross Hospital, London, England
  - University College London Hospitals NHS Foundation Trust, University College Hospital, London, England
  - Salford Royal NHS Foundation Trust, Salford Hospital, Manchester, England
  - Oxford University Hospitals NHS Foundation Trust, John Radcliffe Hospital, Oxford, England
  - University Hospitals Plymouth NHS Trust, Derriford Hospital, Plymouth, England
  - Sheffield Teaching Hospitals, Sheffield, England
  - University Hospitals of North Midlands, Stoke, England
  - Royal Infirmary of Edinburgh, Edinburgh, Scotland
  - Cardiff and Vale University Local Health Board, University Hospital of Wales, Cardiff, Wales
  - Aneurin Bevan Local Health Board Headquarters, Royal Gwent Hospital, Newport, Wales
  - Swansea Bay University Local Health Board, Morriston Hospital, Swansea, Wales
  - Nottingham University Hospitals NHS Trust, Queens Medical Centre, Nottingham

IPD SHARING:
Plan to Share IPD: No